CLINICAL TRIAL: NCT01264796
Title: Community-Based Diabetes Care for Korean American Immigrants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Miyong Kim, Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R18DK083936-01 (NIH); 1R18DK083936-01 (NIH)
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2012-03

CONDITIONS: Type 2 Diabetes
Keywords: Korean American, type 2 diabetes, culturally tailored
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- behavioral intervention, counseling (Experimental): 2hr group education for 6 weeks
  Interventions: Behavioral: culturally tailored diabetes education
- delyed intervention (No Intervention): control group

INTERVENTIONS:
Behavioral: culturally tailored diabetes education — lifestyle modification group education
  Other Names: lifestyle modification
  Arms: behavioral intervention, counseling

SUMMARY:
The primary aims are to test the effectiveness of the self-help DM intervention (SHIP-DM), a comprehensive, culturally tailored DM management intervention, in improving glucose outcomes; To determine the effectiveness of the SHIP-DM in KAI with type 2 DM in improving self-care skills and psycho-behavioral outcomes related to DM control, to develop tangible infrastructures for the dissemination of valid and effective education materials to a wider population of KAI with type 2 DM in the US (e.g., audio-visual education materials, web-based intervention materials, mobile telephone-based intervention materials) and to explore the feasibility and acceptability of each dissemination module, utilizing the delayed intervention group participants. The secondary aims are to obtain preliminary cost-effectiveness data related to the proposed intervention, including cost estimates for this type of DM intervention, and to establish a systematic, long-term dissemination plan, including documenting effective methodologies, to facilitate faster translation of research findings and products to direct consumers in non-research settings.

DETAILED DESCRIPTION:
Inclusion Criteria

1. Self-identified as a first generation Korean American
2. Type 2 diabetes
3. Age 30-75 years
4. Resides in Washington-Baltimore area
5. Self-identified with DM and HbA1c >= 7.0 % within 6 months of screening
6. Expresses willingness to participate in all aspects of the study over its full course

Exclusion criteria

1. Unable to give informed consent
2. Physical or mental health conditions that could limit active participation in the study (e.g., blindness in both eyes, severe immobility, psychiatric diseases)
3. Hematological condition that would affect A1C assay, e.g., hemolytic anemia, sickle cell anemia
4. Past experience in diabetes group education

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified as a first generation Korean American
2. Type 2 diabetes
3. Age 30-75 years
4. Resides in Washington-Baltimore area
5. Self-identified with DM and HbA1c >= 7.0 % within 6 months of screening
6. Expresses willingness to participate in all aspects of the study over its full course

Exclusion Criteria:

1. Unable to give informed consent
2. Physical or mental health conditions that could limit active participation in the study (e.g., blindness in both eyes, severe immobility, psychiatric diseases)
3. Hematological condition that would affect A1C assay, e.g., hemolytic anemia, sickle cell anemia
4. Past experience in diabetes group education

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-11; Primary Completion 2014-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12month
  HbA1c level change from baseline comparing with control group
Blood pressure | 12 month
  BP change from baseline comparing with control group
Lipid profile | 12 months
  LDL level change from baseline comparing with control group
quality of life | 12month
  quality of life score change from baseline comparing with control group

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Kim MT, Kim KB, Ko J, Murry N, Xie B, Radhakrishnan K, Han HR. Health Literacy and Outcomes of a Community-Based Self-Help Intervention: A Case of Korean Americans With Type 2 Diabetes. Nurs Res. 2020 May/Jun;69(3):210-218. doi: 10.1097/NNR.0000000000000409. PMID 31972848
- [Derived] Kim MT, Kim KB, Ko J, Murry N, Levine D, Lee JY. The Differential Role of Vitamin D in Type 2 Diabetes Management and Control in Minority Populations. J Immigr Minor Health. 2019 Dec;21(6):1266-1274. doi: 10.1007/s10903-019-00857-x. PMID 30747313
- [Derived] Kim MT, Kim KB, Ko J, Jang Y, Levine D, Lee HB. Role of depression in diabetes management in an ethnic minority population: a case of Korean Americans with type 2 diabetes. BMJ Open Diabetes Res Care. 2017 Mar 24;5(1):e000337. doi: 10.1136/bmjdrc-2016-000337. eCollection 2017. PMID 28405343
- [Derived] Kim MT, Kim KB, Huh B, Nguyen T, Han HR, Bone LR, Levine D. The Effect of a Community-Based Self-Help Intervention: Korean Americans With Type 2 Diabetes. Am J Prev Med. 2015 Nov;49(5):726-737. doi: 10.1016/j.amepre.2015.04.033. Epub 2015 Jul 14. PMID 26184986